CLINICAL TRIAL: NCT04433182
Title: Copanlisib in Combination With Rituximab-Bendamustine in Patients With Relapsed-Refractory Diffuse Large B-cell Lymphoma: a Multicentric Phase II Trial
Brief Title: Copanlisib With Rituximab-Bendamustine in Patients With Relapsed-Refractory Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_Copa-RB
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse Large B-cell Lymphoma; Relapsed-Refractory; DLBCL; Copanlisib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm Copa-RB (Experimental): Induction phase with Copanlisib, Rituximab and Bendamustina. Maintenance phase (for patients who reach at least SD after induction) with Copanlisib in monotherapy.
  Interventions: Drug: Copanlisib

INTERVENTIONS:
Drug: Copanlisib — Induction phase: 6 cycles of Copa-RB every 28 days according to the following schedule
  * Copanlisib (Copa): 60 mg/day i.v. on days 1,8,15
  * Rituximab (R): 375 mg/sqm i.v. day 1*
  * Bendamustine (B): 90 mg/sqm i.v. days 1-2*
  note: during cycle 1 rituximab can be administered on day 2: in this case bendamustine will be administered on days 2-3; in the case of a frail patient or a patient with high tumor burden copanlisib could be administered on day 1, rituximab on day 2 and bendamustine on days 3-4, at physician discretion.
  Maintenance phase: patients who reach at least SD after induction will receive a maintenance with copanlisib in monotherapy according to the following schedule:
  • Copanlisib: 60 mg/day i.v. on days 1 and 15 in 28-day cycles for 1 year
  Other Names: ALIQOPA

SUMMARY:
This is a multicentric single arm phase II trial, to investigate the efficacy (in terms of PFS) of the combination regimen rituximab-bendamustine in association with copanlisib in patients affected by relapsed/refractory DLBCL, not eligible to HDC and ASCT or relapsed after intensified regimens.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy, in terms of Progression Free Survival (12m-PFS) at 12 months, of a treatment with copanlisib in combination with a standard rituximab-bendamustine regimen in patients with relapsed-refractory DLBCL, who have received at least one, but no more than three lines of treatment, including rituximab-based immunochemotherapy, not eligible for high-dose chemotherapy and ASCT or T-cell CAR-T therapy, or relapsed after these treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of DLBCL (de-novo DLBCL or DLBCL transformed by indolent lymphoma) including:

   * DLBCL, NOS including GCB type, ABC type;
   * T-cell rich large B-cell Lymphoma;
   * Epstein-Barr virus-positive DLBCL, NOS;
   * High-grade B-cell Lymphoma with MYC and BCL2 and/or BCL6 rearrangements (double- hit or triple-hit lymphoma);
   * High-grade B-cell lymphoma NOS;
   * Intravascular B-cell Lymphoma;
   * Extranodal DLBCL;
   * DLBCL coexistent with either follicular lymphoma of any grade or marginal-zone lymphoma;
   * FL grade 3b. Patients must be CD20 positive. New biopsy at relapse time is recommended, but not mandatory.
2. Patients must have relapsed (recurrence after complete response or presented progression after partial response) or refractory after at least ≥ 1 (but < 4) prior lines of therapy, including rituximab-based immunochemotherapy.

   A previous regimen is defined as one of the following: at least 2 months of single-agent therapy; at least 2 consecutive cycles of polychemotherapy; autologous transplant; radioimmunotherapy.
3. Patients must not be eligible to high-dose chemotherapy (HDC) and autologous stem cell transplantation (ASCT) or relapsed after that.
4. Patients must not be eligible to CAR T-cell therapy or relapsed after that.
5. Patients must have at least one bi-dimensionally measurable lesion (that has not been previously irradiated) according to the 2014 Lugano criteria.
6. Male or female patient ≥ 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 if not related to lymphoma disease.
8. Ann Arbor stage II-IV disease.
9. Life expectancy of at least 3 months.
10. Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and 6 months after last administration of bendamustine or copanlisib or 12 months after last rituximab dose. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control method (failure rate of less than 1%) e.g. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.
11. Adequate liver, renal and bone marrow function, assessed by baseline laboratory values as assessed within 7 days before starting study treatment; as assessed by the following (ULN= upper level of normality):

    * Total bilirubin ≤ 1.5 x ULN (< 3 x ULN for patients with Gilbert-Meulengracht syndrome, patients with cholestasis due to compressive adenopathies of the hepatic hilum or documented liver involvement by lymphoma).
    * Alanine transaminase (ALT or GPT) and aspartate aminotransferase (AST or GOT) < 2.5 x ULN (< 5x ULN for patients with documented liver involvement or with biliary obstruction due to lymphoma).
    * Lipase ≤ 1.5 x ULN.
    * Glomerular filtration rate (GFR) ≥ 30mL/min/1.73 m2 according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula. If not on target, this evaluation may be repeated once after at least 24 hours either according to the MDRD abbreviated formula or by 24-hour sampling. If the latter result is within acceptable range, it may be used to fulfil the inclusion criteria instead.
    * International normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 1.5 x ULN. PTT can be used instead of INR if PTT ≤ 1.5 x ULN.
    * Platelet count ≥ 75,000/mm3. For patients with lymphomatous bone marrow infiltration (local assessment) or splenomegaly, platelet count ≥ 50,000/mm3. Platelet transfusion should not be given less than 7 days before the exam collection.
    * Absolute neutrophil count (ANC) ≥ 1,000/mm3 (unless neutropenia related to lymphomatous bone marrow infiltration).
    * Hemoglobin (Hb) ≥ 8 g/dL (unless anemia related to active lymphoma).
12. Left ventricular ejection fraction ≥ 45%.
13. Ability to understand and willingness to sign written informed consent. Signed informed consent must be obtained before any study specific procedure.

Exclusion Criteria:

Patients who meet any of the following criteria at the time of screening will be excluded.

* Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.
* Previous (within 28 days or less than 5 half-lives of the drug before start of study treatment) or concomitant participation in another clinical study with investigational medicinal product(s).

Excluded medical conditions:

1. Primary mediastinal B-cell Lymphoma (PMBCL)
2. DLBCL with concomitant HHV8 positivity or chronic inflammation
3. ALK positive DLBCL
4. Known lymphomatous involvement of the central nervous system
5. Congestive heart failure > New York Heart Association (NYHA) class 2
6. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months).
7. Myocardial infarction less than 6 months before start of test drug
8. Uncontrolled arterial hypertension despite optimal medical management
9. HbA1c> 8.5%
10. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication. Patients with venous thrombotic events related to lymphoma vascular infiltration or compressive disease are eligible providing no signs of pulmonary embolism
11. Non-healing wound, ulcer, or bone fracture
12. Active, clinically serious infections > CTCAE Grade 2
13. History of, or current autoimmune disease
14. Known history of Human immunodeficiency virus (HIV) infection. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations.
15. DLBCL with concomitant primitive or secondary immunodeficiency
16. Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel. Patients positive for HBsAg are excluded. Patients positive for HBcAb will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA
17. CMV PCR positive at baseline
18. Previous or concurrent history of malignancies other than DLBCL within 5 years prior to study treatment except for curatively treated:

    * Cervical carcinoma in situ
    * Non-melanoma skin cancer
    * Superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
    * Localized prostate cancer
19. Patients with seizure disorder requiring medication
20. Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication
21. Proteinuria of ≥ CTCAE Grade 3 as assessed by a 24h protein quantification or estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
22. History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
23. Concurrent diagnosis of pheochromocytoma
24. Pregnant or breast-feeding patients. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.

Patients who meet any of the following criteria at the time of screening will be excluded.

* Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.
* Previous (within 28 days or less than 5 half-lives of the drug before start of study treatment) or concomitant participation in another clinical study with investigational medicinal product(s).

Excluded medical conditions:

1. Primary mediastinal B-cell Lymphoma (PMBCL)
2. DLBCL with concomitant HHV8 positivity or chronic inflammation
3. ALK positive DLBCL
4. Known lymphomatous involvement of the central nervous system
5. Congestive heart failure > New York Heart Association (NYHA) class 2
6. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months).
7. Myocardial infarction less than 6 months before start of test drug
8. Uncontrolled arterial hypertension despite optimal medical management
9. HbA1c> 8.5%
10. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication. Patients with venous thrombotic events related to lymphoma vascular infiltration or compressive disease are eligible providing no signs of pulmonary embolism
11. Non-healing wound, ulcer, or bone fracture
12. Active, clinically serious infections > CTCAE Grade 2
13. History of, or current autoimmune disease
14. Known history of Human immunodeficiency virus (HIV) infection. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations.
15. DLBCL with concomitant primitive or secondary immunodeficiency
16. Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel. Patients positive for HBsAg are excluded. Patients positive for HBcAb will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA
17. CMV PCR positive at baseline
18. Previous or concurrent history of malignancies other than DLBCL within 5 years prior to study treatment except for curatively treated:

    * Cervical carcinoma in situ
    * Non-melanoma skin cancer
    * Superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
    * Localized prostate cancer
19. Patients with seizure disorder requiring medication
20. Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication
21. Proteinuria of ≥ CTCAE Grade 3 as assessed by a 24h protein quantification or estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
22. History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
23. Concurrent diagnosis of pheochromocytoma
24. Pregnant or breast-feeding patients. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
25. Unresolved toxicity higher than CTCAE Grade 1 attributed to any prior therapy/procedure, excluding alopecia
26. Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation
27. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
28. Any illness or medical conditions that are unstable or could jeopardize the safety of patients and their compliance in the study e.g., uncontrolled diabetes, uncontrolled dyslipidemia, etc.)

Excluded previous therapies and medications:

* Prior treatment with copanlisib.
* Prior exposure to idelalisib or other PI3K inhibitors, less than 28 days before start of treatment, unless evidence of progression since last treatment
* Prior treatment with bendamustine: subjects treated with bendamustine at least 24 months before, with a response > one year to bendamustine containing regimen, will be eligible
* Ongoing immunosuppressive therapy.
* Radiotherapy or immuno-/chemotherapy less than 2-4 weeks before start of treatment (corticosteroids are allowed) and use of myeloid growth factors within 14 days prior to treatment
* platelet transfusion less than 7 days before start of treatment
* Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not allowed. Previous corticosteroid therapy must be stopped or reduced to the allowed dose 7 days before performing the screening PET or PET/CT and/or CT/MRI, whichever is performed first, and again prior to the first study drug administration. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose after the patient has signed the IC. Patients may be using topical or inhaled corticosteroids. A pre-phase with corticosteroids is allowed to control the disease in case of systemic symptoms and/or compressive disease with a maximum of prednisone 100 mg (or equivalent) daily for a maximum of 15 days prior start of treatment.
* Autologous transplant less than 2 months before start of treatment. Prior Autologous stem cell performed more than 2 months before start of treatment is allowed.
* History of having received an allogeneic bone marrow or organ transplant.
* Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of treatment or have not recovered from major side effects.
* Anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Use of CYP3A4 inhibitors and inducers. Copanlisib is primarily metabolized by CYP3A4. Therefore, concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted from Day -28 of Cycle 1 until restaging at the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 4 years
  Progression-Free Survival (PFS) will be defined as the time between the date of enrolment and the date of disease progression, relapse or death from any cause. Responding patients according to Response Criteria for NHL with PET and patients who are lost to follow-up will be censored at their last assessment date.

SECONDARY OUTCOMES:
Overall Survival (OS) | 4 years
  Time between the date of enrolment and the date of death from any cause. Patients who have not died at the time of the final analysis will be censored at the date of the last contact.
Overall Response Rate (ORR) | End of treament (EOT), 30 months
  ORR will be defined as the sum of CR + PR
Complete Response Rate (CRR) | End of induction (EOI), 18 months
  CRR will be defined as the proportion of patients achieving a CR
Duration of response (DOR) | 4 years
  DOR is measured from the date when criteria for response are met (CR or PR) until the date of progression or relapse. Patients without relapse or progression will be censored at their last assessment date.
Conversion rate from SD/PR to PR/CR with maintenance | End of treatment (after maintenance), 30 months
  Conversion rate from SD/PR to PR/CR with maintenance
Evaluation of adverse events according to the current version of the CTCAE criteria | 4 years
  Evaluation of adverse events according to the current version of the CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, Principal Investigator — Ematologia, Candiolo Cancer Institute. FPO-IRCCS
Locations (17):
- Italy (17):
  - Ospedale Monsignor Raffaele Dimiccoli - Ematologia, Barletta, Barletta-Andria-Trani
  - Centro Riferimento Oncologico - S.O.C. Oncologia Medica A, Aviano, Pordenone
  - Ematologia, Candiolo Cancer Institute. FPO-IRCCS, Candiolo, Torino
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - ASST Spedali Civili - Ematologia, Brescia
  - Arnas Nuovo Ospedale Garibaldi Nesima - U.O.C. Ematologia, Catania
  - A.O. S. Croce e Carle - S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - Ospedale Vito Fazzi - Ematologia, Lecce
  - Azienda Ospedali Riuniti Papardo-Piemonte - S.C. Ematologia, Messina
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - AOU Policlinico Giaccone - Ematologia, Palermo
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - Azienda Ospedaliera Sant'Andrea - Ematologia, Roma
  - Policlinico Umberto I - Università "La Sapienza" Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Azienda Ospedaliera S. Maria di Terni - S.C. Oncoematologia, Terni
  - Azienda Ospedaliero Universitaria Città della Salute e della Scienza - S.C.Ematologia, Torino
  - Ospedale Ca' Foncello - S.C di Ematologia, Treviso

IPD SHARING:
Plan to Share IPD: No